CLINICAL TRIAL: NCT03892122
Title: Randomised Monocentric -Controlled Study to Evaluate the Efficacy and Stability of Dexmedetomidine Sedation Compared to Propofol Sedation in the Routinely Diagnostic Examination: Drug Induced Sleep Endoscopy
Brief Title: Efficacy and Stability of Dexmedetomidine Sedation Compared to Propofol Sedation in the Drug Induced Sleep Endoscopy
Acronym: DISERT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ospedale Monsignor R. Dimiccoli, Barletta (Other)
Responsible Party: Principal Investigator, Michele Barbara, Director, Head of Otolaryngology, Ospedale Monsignor R. Dimiccoli, Barletta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 01-19; 2019-001429-28 (EudraCT Number)
Record Dates: First submitted 2019-03-22; First posted 2019-03-27 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Drug-induced sleep endoscopy; Dexmedetomidine; Airway collapsibility; Propofol
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: it's a randomized controlled single center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol group (Other): Sleep endoscopy will be performed by a Target Controlled Infusion system (BRAUN perfusion system) using Schneider model in effect-site (cerebral) targeted infusion 50-ml prefilled syringe of 1% propofol. Schneider system is a complex pharmacokinetic/pharmacodynamic (PK/PD) model that allows to obtain different rates of drug from the values of age, height, weight and lean body mass of the patient
  . The starting dose of propofol will be 2-2,5 mcg ml-1 and increments of 0.2 mcg ml-1 took place when the new cerebral concentration of propofol will be reached, and never before 5 minutes. In this way, the investigators will be realized a slow technique of TCI propofol infusion according to European working group
  Interventions: Drug: Propofol Fresenius
- Dexmedetomidine group (Other): For the D-DISE group, dexmedetomidine will be administered with an IV infusion at 1 mcg/kg over 10 minutes, followed by a maintenance rate of 0,7 mcg/kg/h.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol Fresenius — Propofol will be infused with TCI (Target Controlled Infusion) pump. TCI system has been developed to provide improved convenience and control during intravenous anaesthesia. The basic principle is that the anesthetist sets and adjusts the target blood concentration- and depth of anesthesia-as required on clinical grounds.
  Infusion rates are altered automatically according to a validated pharmacokinetic model. TCI technology uses different pharmacokinetic modeling to control the infusion rate of the pump, which allows for a direct control of the sedative agent brain concentration rather than its blood concentration. (de vito 2017) The development of target-controlled infusion (TCI) technology has increased the number of indications for propofol sedation in clinical practice. Furthermore, several studies have demonstrated that propofol-based TCI allows for the accurate control of sedation during DISE and results in an authentic reproduction of the sleep process.
  Arms: Propofol group
Drug: Dexmedetomidine — is a selective alpha-2 adrenergic receptor agonist, which seems to act on the locus coeruleus (LC) or to the preoptic hypothalamus to decrease wakefulness, with almost no effect on respiratory depression. Dexmedetomidine exerts its hypnotic action through activation of central pre- and postsyn¬aptic alpha2-receptors in the locus coeruleus, thereby inducting a state of unconsciousness similar to natural sleep, with the unique as¬pect that patients remain easily arousable and cooperative. Comparing with propofol, dexmedetomidine provides a state of sedation closer to natural sleep and lesser upper airways muscular relaxing effect, even at the increased anesthetic dosage Otherwise, Dexmedetomidine is characterized by a slightly longer onset of action (5-10 minutes), and patients take longer timing to recover..The sedative action of Dexmedetomidine can be reached by means of infusion technique (starting dose: 1 μg/kg over 10 minutes; maintenance infusion rate: 0,7 μg/kg/h).
  Arms: Dexmedetomidine group

SUMMARY:
Obstructive Sleep Apnea Syndrome affect up 12% in adult population. It is associated with an increase rate of hypertension, metabolic syndrome, depression and adverse cardiovascular events. The evaluation of upper airway obstruction is vital to obtain site-specific treatment. Drug Induced Sleep Endoscopy (DISE) is a routinely exam which allows the direct observation of the upper airway during sedative induced sleep. Propofol and Dexmedetomidine are sedatives approved for all diagnostic examinations that required sedation.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea Syndrome affect up 12% in adult population. It is associated with an increase rate of hypertension, metabolic syndrome, depression and adverse cardiovascular events. The evaluation of upper airway obstruction is vital to obtain site-specific treatment. Drug Induced Sleep Endoscopy is a routinely exam which allows the direct observation of the upper airway during sedative induced sleep. Propofol and Dexmedetomidine are sedatives approved for all diagnostic examinations that required sedation.

It's a Randomized Controlled study. 28 participants will be enrolled and randomized in two groups: in the first group the sedation state will be performed with Propofol, while in the second group will be used Dexmedetomidine for allow sedation state. The study will be evaluate the different hemodynamic and respiratory changes during sedation in these two different groups and differences in obstructive endoscopic anatomical patterns. This will be the first study in whic Dexmedetomidine and Propofol will be compared according to European DISE Recommendation published in august 2018 (references)

ELIGIBILITY:
Inclusion Criteria:

* Apnea-Hypopnea Index (AHI) of 15-30.
* Men and women, age 18-65 years, Body Mass Index (BMI) < 35 Kg/m2,
* Awake oxygen saturation > 95%
* Able to read and sign the consent form

Exclusion Criteria:

* Chronic Obstructive Pulmonary Disease (COPD)
* Liver disease (Child Pugh 1-3)
* History of chronic use of sedatives, narcotics, alcohol or illicit drugs,
* History of 1st and 2nd degree heart block (not paced),
* Left Ventricular Ejection Fraction (LVEF) < 50%,
* Allergy to propofol or Dexmedetomidine,
* OSHAS (Obstructive sleep apnea/hypopnea syndrome) surgical failure patients
* Pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-03-22 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
oxygen saturation variation during DISE | during DISE time (until 40 minutes)
  every 5 minute will be recorded this variation and for all exam duration
hert rate variation during DISE | during DISE time (until 40 minutes)
  every 5 minute will be recorded this variation and for all exam duration
systolic and diastolic blood pressure variation during DISE | during DISE time (until 40 minutes)
  every 5 minute will be recorded this variation and for all exam duration
adverse events during DISE | during DISE time (until 40 minutes)
  Number of Participants with arterial hypotension, hypertension; number of desaturation episodes below 60%; rate of patients with heart rate below 50 beats per minute.

SECONDARY OUTCOMES:
pharyngeal and laryngeal patterns during DISE | during DISE time (until 40 minutes)
  pharyngeal and laryngeal patterns observed during DISE will be compared with patterns observed during awake endoscopic evaluation, the vote classification will be used

CONTACTS AND LOCATIONS:
Overall Officials: Michele Barbara, MD, Principal Investigator — Otorhinolaryngology Department of Barletta's hospital; Francesco Barbara, MD, Study Chair — Otorhinolaryngology department of " Policlinico di Bari"; Ilaria Alicino, MD, Study Chair — Anesthesia Department of Barletta's hospital; Valentina Dibenedetto, MD, Study Chair — Otorhinolaryngology Department of Barletta's hospital
Locations (1):
- U.O.C. Otorinolaringoiatria Ospedale Di Barletta, Barletta, BAT, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Padiyara TV, Bansal S, Jain D, Arora S, Gandhi K. Dexmedetomidine versus propofol at different sedation depths during drug-induced sleep endoscopy: A randomized trial. Laryngoscope. 2020 Jan;130(1):257-262. doi: 10.1002/lary.27903. Epub 2019 Mar 1. PMID 30821349
- [Background] Zhao LL, Liu H, Zhang YY, Wei JQ, Han Y, Han L, Yang JP. A Comparative Study on Efficacy and Safety of Propofol versus Dexmedetomidine in Sleep Apnea Patients undergoing Drug-Induced Sleep Endoscopy: A CONSORT-Prospective, Randomized, Controlled Clinical Trial. Biomed Res Int. 2018 Nov 1;2018:8696510. doi: 10.1155/2018/8696510. eCollection 2018. PMID 30515416
- [Background] Viana A, Zhao C, Rosa T, Couto A, Neves DD, Araujo-Melo MH, Capasso R. The Effect of Sedating Agents on Drug-Induced Sleep Endoscopy Findings. Laryngoscope. 2019 Feb;129(2):506-513. doi: 10.1002/lary.27298. Epub 2018 Sep 7. PMID 30194726
- [Background] De Vito A, Carrasco Llatas M, Ravesloot MJ, Kotecha B, De Vries N, Hamans E, Maurer J, Bosi M, Blumen M, Heiser C, Herzog M, Montevecchi F, Corso RM, Braghiroli A, Gobbi R, Vroegop A, Vonk PE, Hohenhorst W, Piccin O, Sorrenti G, Vanderveken OM, Vicini C. European position paper on drug-induced sleep endoscopy: 2017 Update. Clin Otolaryngol. 2018 Dec;43(6):1541-1552. doi: 10.1111/coa.13213. Epub 2018 Sep 30. PMID 30133943
- [Background] De Vito A, Agnoletti V, Zani G, Corso RM, D'Agostino G, Firinu E, Marchi C, Hsu YS, Maitan S, Vicini C. The importance of drug-induced sedation endoscopy (D.I.S.E.) techniques in surgical decision making: conventional versus target controlled infusion techniques-a prospective randomized controlled study and a retrospective surgical outcomes analysis. Eur Arch Otorhinolaryngol. 2017 May;274(5):2307-2317. doi: 10.1007/s00405-016-4447-x. Epub 2017 Feb 17. PMID 28213776
- [Background] De Vito A, Agnoletti V, Berrettini S, Piraccini E, Criscuolo A, Corso R, Campanini A, Gambale G, Vicini C. Drug-induced sleep endoscopy: conventional versus target controlled infusion techniques--a randomized controlled study. Eur Arch Otorhinolaryngol. 2011 Mar;268(3):457-62. doi: 10.1007/s00405-010-1376-y. Epub 2010 Sep 2. PMID 20811901